CLINICAL TRIAL: NCT00902148
Title: Evaluation of Intra-Abdominal Adhesions in Ileostomy Procedures When Using a Resorbable Polylactide Film (SurgiWrap) in Colorectal Surgeries
Brief Title: Evaluation of Bioresorbable Sheet to Prevent Intra-Abdominal Adhesions in Colorectal Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MAST Biosurgery, AG (Industry)
Responsible Party: Arne E. Faerden, MD, Akershus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20031124
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Adhesions
Keywords: Surgery; Colectomy; Proctocolectomy; Adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Colorectal Surgery without use of SurgiWrapTM
- Test Group (Active Comparator): Colorectal Surgery with use of SurgiWrapTM film secured directly below the abdominal incision
  Interventions: Device: Polylactic Acid Sheet

INTERVENTIONS:
Device: Polylactic Acid Sheet — SurgiWrapTM bioresorbable sheet will be secured directly below the abdominal incision.
  Other Names: SurgiWrapTM
  Arms: Test Group

SUMMARY:
Study to investigate and determine the difference between the extent and severity of intra-abdominal adhesions in patients where SurgiWrap film was placed compared to patients with no adhesion barrier inserted.

Hypothesis: Due to the preclinical safety data and clinical case reports in various indications it is anticipated that the surgical sites where the resorbable anti-adhesion barrier SurgiWrap was placed, there will be a reduction of adhesions compared to the control group with no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer, ulcerative colitis or other pathologies requiring a second surgery for ileostomy closure.
* Age between 18 and 78 years.
* Patient or his/her legal representative has read and signed the approved Informed Consent form before randomization.

Exclusion Criteria:

* Previous abdominal operation through a midline approach
* Use of hernia mesh
* Use of any antiadhesive irrigants or irrigants containing corticosteroids, heparin, salicylates, nonsteroidal anti-inflammatory drugs.
* Pregnancy

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Assess the extent and severity of new formed adhesions having its source in the target region where the SurgiWrap film initially was placed: between the midline incision/scar and the omentum, and between the midline incision/scar and the small bowel | 6 to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Arne Faerden, MD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Oslo County, Norway